CLINICAL TRIAL: NCT05405062
Title: Efficacy of Carboxytherapy Versus Short-pulsed 1064 nm Nd-YAG Laser Combined With Subcision in Treatment of Cellulite
Brief Title: Carboxytherapy Versus Short-pulsed Nd Yag Laser in Cellulite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carboxy therapy and cellulite
Record Dates: First submitted 2022-01-07; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Efficacy of Treatment of Cellulite Using Carboxy Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carboxytherapy (Active Comparator): Six carboxytherapy sessions with an interval of 2 weeks. Five ccs will be injected at each point with a depth of 7mm. Between each point and the other is 5 cm.
  Interventions: Device: Carboxytherapy, short pulsed 1064 Nd Yag laser and subcision
- Short pulsed 1064 nm Nd-YAG laser combined with subcision (Active Comparator): Twenty-five joules/cm2, 2.2Hz combined with subcision with an interval of 1 month.
  Interventions: Device: Carboxytherapy, short pulsed 1064 Nd Yag laser and subcision

INTERVENTIONS:
Device: Carboxytherapy, short pulsed 1064 Nd Yag laser and subcision — Carboxytherapy is involves the injection of carbon dioxide into the subcutaneous tissue, with the goal of affecting the adipose tissue and circulation. Its mechanism of action is through an increase in capillary blood flow induced by hypercapnia and a decrease in cutaneous oxygen consumption (Pianez et al., 2016).

SUMMARY:
To evaluate the efficacy of carboxytherapy versus short-pulsed 1064 nm Nd-YAG laser combined with subcision in treatment of cellulite using clinical assessment and ultrasound imaging.

DETAILED DESCRIPTION:
Study Design:

Randomized Clinical Trial

Study Methods:

The population of study: Thirty females aged from 18 to 60 years with cellulite Study location: Dermatology outpatient clinic, Faculty of Medicine, Cairo University

Inclusion criteria:

1. Females between 18 and 60 years
2. Females with cellulite; stage 2 or 3 according to Nurnberger-Muller Scale

Exclusion criteria:

1. Subjects that have had liposuction or surgical procedures to remove fat in the past 6 months
2. Personal or family history of keloid formation or scarring
3. Pregnant or lactating females
4. Significant concomitant illness (e.g. renal, cardiac, hepatic, autoimmune conditions)
5. Known history of bleeding tendency or receiving antiplatelet or anticoagulant therapy
6. History of uncontrolled diabetes
7. History of thrombophlebitis within the last 2 years
8. Subjects with active infections
9. Subjects on long term corticosteroid or immunosuppressive therapy

All patients will be subjected to the following:

An informed written consent will be obtained from all the patients.

* Patients will be examined to assess site, stage and severity of cellulite.
* Depressed areas on gluteal region and posterolateral thighs will be selected and marked while the patient is standing.
* One side will be randomized to receive 6 carboxytherapy sessions with an interval of 2 weeks.
* The other side will receive 3 sessions of short pulsed 1064 nm Nd-YAG laser (25 joules/cm2, 2.2Hz) combined with subcision with an interval of 1 month.
* In carboxytherapy, 5 cc will be injected in each point with depth of 7mm. Between each point and the other is 5 cm.
* Subcision will be done in the center of the selected dimples.
* Systemic antibiotics will be prescribed for 5 days after subcision session.
* The whole duration of the sessions is 3 months.
* Patients will be advised to maintain a healthy diet throughout the study.

Evaluation of patients' response:

* A complete physical examination and history taking before treatment
* Evaluation will be carried out for each patient at the beginning of the study, and at the end of the study 2 weeks following the final session by:

  1. Standardized photography (posterior and side view)
  2. Photonumeric cellulite severity scale (Hexsel et al., 2009)
  3. Ultrasound imaging that measures percentage of reduction of subcutaneous fat and dermal thickness. The device used is Toshiba with high frequency probes: probe 18-20 MHz (for measuring skin dermal thickness) and probe 7-9MHz (for measuring subcutaneous fat thickness)
  4. Patient satisfaction scoring will be reported at the end of the study by patient satisfaction score (excellent, very good, good, bad, very bad) and DLQI score (Finlay and Khan, 1994).

Potential risks:

1. Ecchymosis
2. Pain
3. Burning sensation

3- Secondary infection at injection site

Study outcomes:

1. Assessment of efficacy of carboxytherapy in the treatment of cellulite (clinically by photography and photonumeric severity scale).
2. Evaluating possible synergistic effect of short pulsed Nd-YAG laser combined with subcision in treatment of cellulite (clinically by photography and photonumeric severity scale).

Secondary outcome:

Comparing the reduction in subcutaneous fat and change in dermal thickness between the 2 methods by ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 18 and 60 years
2. Females with cellulite; stage 2 or 3 according to Nurnberger-Muller Scale (Nurnberger and Muller, 1978)

Exclusion Criteria:

1. Subjects that have had liposuction or surgical procedures to remove fat in the past 6 months
2. Personal or family history of keloid formation or scarring
3. Pregnant or lactating females
4. Significant concomitant illness (e.g. renal, cardiac, hepatic, autoimmune conditions)
5. Known history of bleeding tendency or receiving antiplatelet or anticoagulant therapy
6. History of uncontrolled diabetes
7. History of thrombophlebitis within the last 2 years
8. Subjects with active infections
9. Subjects on long term corticosteroid or immunosuppressive therapy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Photonumeric cellulite severity scale | Change from baseline at 3 months

SECONDARY OUTCOMES:
Ultrasound imaging | Change from baseline at 3 months
  The device used is Toshiba with high frequency probes: probe 18-20 MHz (for measuring skin dermal thickness) and probe 7-9MHz (for measuring subcutaneous fat thickness)